CLINICAL TRIAL: NCT06284096
Title: Effect Of CHIME Based Group Psychoeducation On Personel Recovery In Individuals Diagnosed With Schizophrenia
Brief Title: The Personal Recovery Based Psychoeducation For Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gülnur Sahin, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/391
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Mental Health Recovery; Schizophrenia
Keywords: personal recovery; schizophrenia; wellbeing; CHIME
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group, on the other hand, is aimed at participating in both the psychoeducation program conducted by the researcher and these routine practices within the institution.
  Interventions: Behavioral: Psychoeducation
- Control Group (No Intervention): The control group is planned to participate only in the routine Community Mental Health Center activities within the institution, such as handicraft activities, art, music, computer courses, etc.

INTERVENTIONS:
Behavioral: Psychoeducation — The study is planned to consist of 7 sessions, occurring once a week, with approximately 60-70 minutes allocated for each session. Considering the attention span of the participants, the sessions will be divided into two parts, with a session lasting 30-40 minutes followed by a 15-minute break.
  Arms: Intervention group

SUMMARY:
This project aims to introduce a new psychoeducation program that helps individuals with schizophrenia to recover subjectively. The program's effectiveness will be evaluated through a randomized controlled research design. The goal is not only to emphasize clinical recovery but also to highlight the importance of individual recovery and promote its implementation. In this context, the following hypotheses have been formulated.

Research Question:

1) Does recovery-based psychoeducation have an impact on the subjective recovery level in individuals diagnosed with schizophrenia in remission?

Hypotheses:

H0a: Recovery-based psychoeducation does not affect the subjective recovery level in individuals diagnosed with schizophrenia in remission.

H0b: Recovery-based psychoeducation does not effect on psychological resilience in individuals diagnosed with schizophrenia in remission.

H0c: Recovery-based psychoeducation does not effect on hope in individuals diagnosed with schizophrenia in remission.

H1a: Recovery-based psychoeducation affects the subjective recovery level in individuals diagnosed with schizophrenia in remission.

H1b: Recovery-based psychoeducation has an effect on psychological resilience in individuals diagnosed with schizophrenia in remission.

H1c: Recovery-based psychoeducation has an effect on hope in individuals diagnosed with schizophrenia in remission.

DETAILED DESCRIPTION:
CHIME (Connectedness-Hope-Identity-Meaning of Life-Empowerment) is a framework conceptualizing subjective recovery in individuals with mental disorders. Based on a systematic review involving 97 studies, five fundamental principles of recovery were identified in these studies. These principles are listed as Empowerment, Hope and Optimism, Connectedness (Social Support), Meaning of Life, and Identity. A psychoeducation program has been developed based on this framework. A study examining 115 international English articles conceptualizing personal recovery revealed that most articles reflected all five recovery components, supporting its validity. In another study evaluating the components of subjective recovery, it was found that most components were necessary for the recovery journey of individuals with different psychiatric diagnoses such as bipolar disorder and eating disorders. Consequently, the recovery framework has gained more importance recently for researchers and clinicians by providing an inclusive consensus model.

The psychoeducation program planned based on the Concept of Personal Recovery aims to accelerate recovery, make it sustainable, and demonstrate the importance of individualized care based on the individual's values and treatment preferences.

Research Design: Pretest-posttest randomized controlled intervention study Population and Sample of the Study: The population of the study consists of 236 individuals diagnosed with schizophrenia, registered at the Umraniye Community Mental Health Center affiliated with Erenkoy Mental and Neurological Diseases Training and Research Hospital, who meet the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria.

To calculate the sample for the study, a preliminary study will be conducted with a group of 10 individuals. Based on the data obtained from this preliminary study, the sample size will be calculated using the G-power program.

Location and Timing of the Research: Approval document with the number 2023/391 from Istanbul University-Cerrahpasa Social and Humanities Research Ethics Committee is available. The data collection and group sessions for the study, scheduled to be conducted between April and June 2024, after obtaining approval from the Ministry of Health, Istanbul Provincial Health Directorate, will take place in the Umraniye Community Mental Health Center meeting room. The meeting room has been designated as a suitable environment for group sessions with the necessary size, no entry or exit during sessions, and conditions suitable for interaction and sharing in terms of safety. In addition, a blackboard and a projector are available for use during the sessions. Group members will be invited on session days within the time frame determined by common agreement.

Data Collection Method:

Data will be collected through the participants filling out the scale with the assistance of a research assistant.

Data Collection Instruments:

Personal Data Form: A form created by the researcher in accordance with the literature, consisting of a total of 9 questions about participants' socio-demographic characteristics and disease conditions.

Subjective Recovery Assessment Scale: A self-report scale developed by Yildiz and colleagues to assess the subjective recovery status of individuals diagnosed with schizophrenia. The scale is a five-point Likert scale, and each item is scored from one to five. An increase in the score indicates that the individual perceives themselves as improved. The scale is evaluated as a single-factor scale without sub-dimensions Psychological Resilience Assessment Scale: Developed by Johnson and colleagues and validated with individuals with mental disorders by Duran. It is a five-point Likert scale consisting of a total of 12 items and two sub-dimensions. These sub-dimensions are named "Social Support" and "Emotional Coping/Situational Coping".

Schizophrenia Hope Scale: Developed by Choe to determine the hope levels of individuals diagnosed with schizophrenia. It consists of a total of 9 questions and has a 3-point Likert-type rating (0=disagree, 1=agree, 2=strongly agree). The total score obtained from the scale ranges from 0 to 18. The scale does not have a cutoff point, and a high score on the scale indicates high hope in individuals diagnosed with schizophrenia. The Turkish validity and reliability study of the scale was conducted by Sahin Altun and colleagues.

Data Collection Tool Implementation and Interventions: Participants who meet the research criteria and agree to participate in the study will be randomized and divided into intervention and control groups. Initial measurements (Personal Data Form, Subjective Recovery Assessment Scale, Psychological Resilience Assessment Scale, Schizophrenia Hope Scale) will be collected by the researcher through face-to-face interviews. While the control group continues to receive routine Community Mental Health Center (CMHC), the intervention group will receive a recovery-oriented psychoeducation program in addition to routine Community Mental Health Center. After the intervention program is completed, the final measurements of both the intervention and control groups will be collected Intervention Stage: It is planned for the control group to participate only in routine Community Mental Health Center activities (craft activities, art, music, computer courses, etc.). The intervention group is aimed to participate in both the psychoeducation program conducted by the researcher and these routine activities in the institution. Interventions will be implemented by the researcher personally. At the end of the intervention, participants will be given an "education evaluation form." The control group will continue with the routine rehabilitation activities implemented at CMHC during this period. The initial meeting with the control group will involve introductions and pre-testing (attachments...abbreviations...). The final testing will be conducted at the end of the period when the intervention group completes the program.

Development of the CHIME Based Group Psychoeducation Program: The program, prepared by the researcher based on relevant literature, has been presented to experts for their opinions. Psychoeducation programs for individuals diagnosed with schizophrenia in the literature have been determined to consist of 5-10 sessions. This study plans to have a total of seven sessions, conducted weekly, with approximately 60-70 minutes allocated for each session, taking into account the attention span of the participants. Sessions will be divided into two parts, each lasting 30-35 minutes with a 15 minute break.

Individuals who voluntarily agree to participate in psychoeducation sessions will be provided with verbal and written consent regarding the group rules. The group rules will be collaboratively determined with the participants. One day before each psychoeducation session, participants will be reminded of the start time through a phone call. Before each session, participants will be supplied with materials such as pens, erasers, and notebooks that they may need and use during the session. To ensure the participants' consistent attendance, the instructor will provide snacks and beverages during each session break.

Session 1: Introduction Introduction of participants to the educator and each other, Purpose, duration, and frequency of the education, Group rules,

Session 2: Identity Rebuilding/redefining positive identity, Overcoming stigma,

Session 3: Meaningful Life Meaning of the mental illness experience, Spirituality, Quality of life, Social roles/goals, Rebuilding life,

Session 4: Hope and Optimism Belief in the possibility of recovery, Motivation for change, Relationships that provide hope,

Session 5: Empowerment Self-management, Control over life, Focusing on strengths,

Session 6: Social Support Peer support and support groups, Friendship relationships, Being a part of the community

Session 7: Process, Evaluation and Closure Reinforcing what has been learned, Program evaluation, Receiving feedback, Certificate, Application of Post-test Measurements.

Scope validity of the Psychoeducation Program: All items of the session content aimed at ensuring the scope validity of the psychoeducation program, prepared in accordance with the relevant literature, were presented to a total of 5 experts who are faculty members in the psychiatry and nursing departments. A scoring form for all session steps was sent to the experts, and they were asked to evaluate the appropriateness of the items in terms of language/culture and content. In the evaluation of expert opinions, Davis' Content Validity Index (CVI) was used. According to the CVI, items receiving 1 and 2 points are unacceptable, and items receiving 3-4 points are considered acceptable. In the analysis, the content validity of the second session (Identity) was calculated as 83%, and the content validity of the other sessions was calculated as 100%, indicating that the psychoeducation has sufficient scope validity.

Randomization: The allocation of individuals included in the study to groups will be determined using a simple random sampling method through www.randomizer.org.

Protection of Participant Confidentiality: During the pre-test and post-test application, participants will be asked to write their initials and the last two digits of their birth year instead of their full names.

Data Analysis: The collected data will be analyzed using the Statistical Package for the Social Sciences Statistics for Windows 20.0 Package. Descriptive analyses, including counts, percentages, means, standard deviations, medians, 25th and 75th percentiles, minimum, and maximum values, will be conducted. The normal distribution of continuous variables will be checked using the Kolmogorov-Smirnov test, and the significance between groups will be compared using parametric tests for those with normal distribution and non-parametric tests for those without normal distribution.

Repeated measures analysis of variance (ANOVA) will be used for the pre-test-post-test evaluation. The comparison of categorical variables will be done using Chi-square tests, and the relationship between variables will be explored using Pearson correlation tests for continuous variables and Spearman correlation tests for discrete variables. Regression analyses will be employed to investigate the impact of independent variables on dependent variables. The statistical significance level in the analyses will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia,
2. Age between 18 and 65,
3. Willingness to participate in the study,
4. At least 6 months in remission,
5. Literacy,
6. No hearing or comprehension problems.

Exclusion Criteria:

1. History of alcohol or substance abuse (excluding nicotine),
2. Presence of comorbid neurocognitive disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Subjective Recovery Assessment Scale | From randomization to end of intervention, in 7 weeks.
  Subjective Recovery Assessment Scale: A self-report scale assess the subjective recovery status of individuals diagnosed with schizophrenia. The scale is a five-point Likert scale, and each item is scored from 1 to 5. An increase in the score indicates that the individual perceives themselves as improved. The scale is evaluated as a single-factor scale without sub-dimensions

SECONDARY OUTCOMES:
Psychological Resilience Assessment Scale | From randomization to end of intervention, in 7 weeks.
  Psychological Resilience Assessment Scale is a five-point Likert scale consisting of a total of 12 items and 2 sub-dimensions. These sub-dimensions are named "Social Support" and "Emotional Coping/Situational Coping. The overall Cronbach's alpha coefficient of the scale was reported as 0.88. The scale does not include any reverse-coded items. The total score of the scale ranges from a minimum of 12 to a maximum of 60. Higher scores indicate higher levels of psychological resilience.
Schizophrenia Hope Scale | From randomization to end of intervention, in 7 weeks.
  Schizophrenia Hope Scale determine the hope levels of individuals diagnosed with schizophrenia. It consists of a total of 9 questions and has a 3-point Likert-type rating (0=disagree, 1=agree, 2=strongly agree). The total score obtained from the scale ranges from 0 to 18. The scale does not have a cutoff point, and a high score on the scale indicates high hope in individuals diagnosed with schizophrenia.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Sukut, Asst. Prof, Study Director — Istanbul University-Cerrahpasa, Florence Nightingale Faculty Of Nursing, Department Of Nursing
Locations (1):
- Umraniye Community Mental Health Center affiliated with the Ministry of Health., Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liberman RP (2009) Recovery from Disability:Manual of Psychiatric Rehabilitation. Washington, American Psychiatric Publication.
- [Background] - Bora S, 2021. The impact of psychoeducation grounded in the Uncertainty in Illness Theory on the uncertainty intolerance, psychological well-being, and coping levels of caregivers providing care to schizophrenia patients. Doctoral Dissertation, Nursing Department, Institute of Health Sciences, Akdeniz University.
- [Background] - Fırıncıoğulları A, 2020. Evaluation of the quality of life and functionality of patients with bipolar disorder after psychoeducation / Mustafa Kemal University, Faculty of Medicine, Department of Psychiatry, Medical Specialization Thesis.
- [Background] - Duran F, 2021. The Relationship between Psychological Resilience, Hopelessness, and Suicidal Thoughts in Adults Diagnosed with Schizophrenia. Master's Thesis, Department of Mental Health Nursing, Istanbul University Cerrahpasa
- [Background] - Ercan Doğu S, 2019. A comparison of the effectiveness of occupational therapy and social skills training in individuals with schizophrenia. Doctoral Dissertation, Hacettepe University, Ankara.
- [Background] - Abaoğlu H, 2018. Investigation of the impact of life skills training on functionality in individuals with schizophrenia. Doctoral Dissertation, Hacettepe University, Ankara.
- [Background] Duval M, Harscoet YA, Jupille J, Grall-Bronnec M, Moret L, Chirio-Espitalier M. Patients' perspectives of the effects of a group-based therapeutic patient education program for bipolar disorder: a qualitative analysis. BMC Psychiatry. 2022 Sep 23;22(1):626. doi: 10.1186/s12888-022-04241-2. PMID 36151517
- [Background] Slade M, Leamy M, Bacon F, Janosik M, Le Boutillier C, Williams J, Bird V. International differences in understanding recovery: systematic review. Epidemiol Psychiatr Sci. 2012 Dec;21(4):353-64. doi: 10.1017/S2045796012000133. Epub 2012 Mar 15. PMID 22794507
- [Background] Shanley E, Jubb-Shanley M. The recovery alliance theory of mental health nursing. J Psychiatr Ment Health Nurs. 2007 Dec;14(8):734-43. doi: 10.1111/j.1365-2850.2007.01179.x. PMID 18039296
- [Background] Wetzler S, Hackmann C, Peryer G, Clayman K, Friedman D, Saffran K, Silver J, Swarbrick M, Magill E, van Furth EF, Pike KM. A framework to conceptualize personal recovery from eating disorders: A systematic review and qualitative meta-synthesis of perspectives from individuals with lived experience. Int J Eat Disord. 2020 Aug;53(8):1188-1203. doi: 10.1002/eat.23260. Epub 2020 Mar 17. PMID 32181532
- [Background] Leamy M, Bird V, Le Boutillier C, Williams J, Slade M. Conceptual framework for personal recovery in mental health: systematic review and narrative synthesis. Br J Psychiatry. 2011 Dec;199(6):445-52. doi: 10.1192/bjp.bp.110.083733. PMID 22130746
- [Derived] Sahin G, Sukut O. Effect of Chime Based Group Psychoeducation on Personal Recovery in Individuals Diagnosed With Schizophrenia. Community Ment Health J. 2025 Nov 15. doi: 10.1007/s10597-025-01555-9. Online ahead of print. PMID 41240240
- See also: A New Direction to Psychiatric Wellness: Recovery Oriented Approach — https://dergipark.org.tr/tr/download/article-file/707300
- See also: Mental Disorder and Recovery — https://doi.org/10.14744/phd.2017.49469
- See also: International differences in understanding recovery: systematic review — https://doi.org/10.1017/S2045796012000133
- See also: Development and preliminary testing of the Schizophrenia Hope Scale, a brief scale to measure hope in people with schizophrenia — https://doi.org/10.1016/j.ijnurstu.2013.10.018
- See also: Conceptual framework for personal recovery in mental health: systematic review and narrative synthesis — http://doi.org/10.1016/j.brat.2009.10.007
- See also: Development and validation of the Subjective Recovery Assessment Scale for patients with schizophrenia — https://doi.org/10.1080/24750573.2017.1405579
- See also: The effect of psychosocial skills training and metacognitive training on social and cognitive functioning in schizophrenia — https://doi.org/10.29399/npa.23095